CLINICAL TRIAL: NCT01601600
Title: A Randomized, Double-blind, Placebo-controlled Multi-center Study to Assess the Effects of BYM338 on Skeletal Muscle in Sarcopenic Adults With Mobility Limitations
Brief Title: A Multi-center Study to Assess the Effects of BYM338 on Skeletal Muscle in Sarcopenic Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBYM338X2201
Record Dates: First submitted 2012-02-17; First posted 2012-05-18 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-11

CONDITIONS: Skeletal Muscle
MeSH Terms: interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BYM338 (Experimental): BYM338 active drug
  Interventions: Drug: BYM338

INTERVENTIONS:
Drug: BYM338 — BYM338
  Arms: BYM338
Drug: Placebo — BYM338 Placebo
  Arms: Placebo

SUMMARY:
The purpose of this Proof of Concept study is to determine the effects of BYM338 on skeletal muscle volume, mass, and strength and patient function (gait speed) in non-demented elderly adults with sarcopenia and mobility limitations. In addition, this study will generate data on the safety, tolerability, and pharmacokinetics of BYM338 in older adults and its response on additional physical function measures in this population. Furthermore, the extended study duration will provide information on the stability of BYM-induced changes in skeletal muscle and patient function in this subgroup of the older population.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 65 or older with difficulty standing up from a chair or walking for longer than 10 minutes on a flat surface or climbing a flight of stairs.
2. Written informed consent must be obtained before any laboratory or physical assessment is performed to establish eligibility. Answering initial questions for qualification, whether in person or over the phone does not require written consent.
3. At the onsite screening, candidates should have gait speed measured over 4 meters of <1.0 m/s but ≥0.6 m/s.
4. Appendicular skeletal muscle index (skeletal muscle in kg/ height in m2) by DXA ≤ 7.25 kg/m2 for men and ≤ 5.67 kg/m2 for women to be assessed during screening if the gait speed criterion in #3 is met.
5. At screening and baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the supine position followed by assessment in standing within three (3) minutes of changing position. Investigators can be guided by the following ranges for the supine measurement and position change:

   * oral body temperature between 35.0-37.5 °C
   * systolic blood pressure, 80-160 mm Hg and a reduction of >20mmHg
   * diastolic blood pressure, 50-90 mm Hg and a reduction of >10mmHg
   * pulse rate, 50 - 100 bpm
6. Patients must weigh at least 35 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 32 kg/m2, inclusive. (See Appendix 4) of this protocol for BMI ranges.
7. Be able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 halflives of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
2. History of hypersensitivity to antibodies.
3. A history of clinically significant ECG abnormalities, which, in the opinion of the investigator, may indicate active cardiac disease.
4. History of malignancy of any organ system (other than localized nonmelanomatous cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
5. Diseases other than cancer known to cause cachexia or muscle atrophy, including but not limited to congestive heart failure of any stage, COPD, chronic kidney disease (estimated GFR < 30 mL/min using the MDRD equation), rheumatoid arthritis, primary myopathy, stroke, HIV infection, tuberculosis or other chronic infection, uncontrolled diabetes mellitus.
6. Diseases known to cause malabsorption of protein or energy, including inflammatory bowel disease, celiac disease, short bowel syndrome, pancreatic insufficiency, etc.
7. Liver disease or liver injury as indicated by abnormal liver function tests such as SGOT (AST), SGPT (ALT), γ-GT, alkaline phosphatase, or serum bilirubin (except Gilbert's

Disease). The Investigator should be guided by the following criteria:

* Any single transaminase listed above may not exceed 3x upper limit of normal (ULN).
* If the total bilirubin concentration is increased above 1.5 x ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed the value of 1.6 mg/dL (27 μmol/L). 8. Use of any prescription drugs known to affect muscle mass, including androgen supplements, anti-androgens (such as LHRH agonists), anti-estrogens (tamoxifen, etc.) recombinant human growth hormone (rhGH), insulin, oral beta agonists, megestrol acetate, dronabinol, etc. 9. Donation or loss of 400 mL or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation. 10. Plasma donation (> 250 mL) within 14 days prior to first dosing. 11. Hemoglobin concentration below 11.0 g/dL at screening. 12. Significant illness within two (2) weeks prior to initial dosing. 13. Patients with known claustrophobia, presence of pacemaker and/or ferromagnetic material in their body that would prohibit administration of MRI assessments. 14. Patient smokes more than one cigarette, pipe or cigar a month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
muscle volume of the thigh (measurement gathered using MRI, magnetic resonance imaging) | baseline to 24 weeks

SECONDARY OUTCOMES:
Safety and tolerability will be measured by physical examination, checking vital signs, ECG evaluation and taking standard laboratory tests. Clinical safety data will be compiled by Adverse events reports. | 24 weeks
Pharmacokinetic profile will measure the (Composite of Pharmacokinetics)area under curve (AUC) | pre-dose, 2, 6 hrs postdose, 1,2,4,6,8,10,12,16,20,40 weeks postdose
Muscle function measured by evaluating physical performance tests | 24 weeks
Health status measured by evaluating patient reports. | 24 weeks
Duration of drug-induced changes in body composition | 24 hours
Duration of drug-induced physical function | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Brighton, Massachusetts

REFERENCES:
- See also: Results for CBYM338X2201 from the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13323